CLINICAL TRIAL: NCT00620997
Title: Challenging the Dogma: Topical Proparacaine is Safe and Effective for the Emergency Department Management of Acute Traumatic Corneal Injuries
Brief Title: Proparacaine vs Placebo for Corneal Injuries
Acronym: Dogma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Dr. Scott Anderson, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: London HSC
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2006-09

CONDITIONS: Corneal Abrasions
Keywords: cornea; analgesia; topical; anesthetic
MeSH Terms: conditions — Corneal Injuries; Corneal Diseases; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients randomized to 0.05% Proparacaine drops on a PRN basis for up to 7 days
  Acetaminophen with Codeine for breakthrough pain
  topical Gatifloxacin drops
  Interventions: Drug: Proparacaine drops 0.05%
- 2 (Placebo Comparator): placebo drops on a PRN basis for up to 7 days post injury
  Acetaminophen with Codeine for breakthrough pain
  Gatifloxacin drops
  Interventions: Drug: saline drops

INTERVENTIONS:
Drug: Proparacaine drops 0.05% — topical, 0.05% drops, PRN continuously for up to 7 days
  Arms: 1
Drug: saline drops — saline drops continuously PRN for up to 7 days
  Arms: 2

SUMMARY:
Introduction: Traumatic injuries to the outer covering of the eye (the cornea) are a common emergency department complaint. They cause significant patient distress including pain, loss of sleep and missed work days. There is currently no accepted, uniform approach to pain management in this patient population. Emergency medicine and ophthalmology texts state that prolonged use of medications that anesthetize the cornea is not recommended. Several recent publications in the ophthalmology literature show that the outpatient use of dilute local anesthesia in patients after eye surgery is a safe and effective method of pain control. In this study, we used Proparacaine (a local anesthetic), in a similar manner, for the outpatient emergency department management of traumatic corneal injuries.

Methods: We performed a clinical trial on a sample of adult patients presenting with traumatic corneal injuries to two university affiliated emergency departments in London, Canada.

Patients providing signed informed consent to participate in the study received a vial of clear liquid that contained either Proparacaine or plain water (placebo), a pain log, topical antibiotics and oral Acetaminophen (Tylenol) with Codeine for breakthrough pain.

Patients were instructed to use the "study drug" on an "as-needed" basis for the next seven days. Patients completed a pain scale describing their discomfort immediately prior to, and five minutes after self-administration of the study drug. All patients were followed closely in an ophthalmology outpatient clinic on Days 1, 3 and 5 after presentation to the emergency department. At the last ophthalmology clinic visit, the patients' pain logs were collected.

The protocol was approved by the Research Ethics Board for Health Sciences Research Involving Human Subjects at the University of Western Ontario.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with acute (within 24 hrs) traumatic corneal injuries

Exclusion Criteria:

* immunocompromised
* known allergy to local anesthetic
* unable to consent /follow instructions for dosing / go to follow-up appointments
* previous ocular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
pain reduction | continuous

SECONDARY OUTCOMES:
patient satisfaction | at 5 days post injury
delayed wound healing | days 3,5 ,7 postinjury

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Anderson, MD FRCPC, Principal Investigator — London Health Sciences Center
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Algarni AM, Guyatt GH, Turner A, Alamri S. Antibiotic prophylaxis for corneal abrasion. Cochrane Database Syst Rev. 2022 May 27;5(5):CD014617. doi: 10.1002/14651858.CD014617.pub2. PMID 35622535